CLINICAL TRIAL: NCT00692640
Title: A Phase 1 Dose-Escalation Study of XL147 (SAR245408) in Combination With Erlotinib in Subjects With Solid Tumors
Brief Title: Safety Study of XL147 (SAR245408) in Combination With Erlotinib in Adults With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED11434; XL147-002 (Other: Other study code)
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Cancer; Non-small Cell Lung Cancer
Keywords: Cancer; Solid Tumors; NSCLC
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — XL147; Erlotinib Hydrochloride

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: XL147 (SAR245408); Drug: Erlotinib

INTERVENTIONS:
Drug: XL147 (SAR245408) — Gelatin capsules supplied in 25-mg and 100-mg strengths; daily dosing for 21 days/7 days off
Drug: Erlotinib — Tablets supplied in 25-mg, 100-mg, and 150-mg strengths; daily dosing
  Other Names: Tarceva®

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of XL147 in combination with erlotinib (Tarceva®) in subjects with solid tumors. XL147 is a new chemical entity that inhibits PI3 Kinase. Inactivation of PI3K has been shown to inhibit growth and induce apoptosis (programmed cell death) in tumor cells. Erlotinib is an orally administered inhibitor of EGFR (also known as HER1) tyrosine kinase. It was approved by the FDA as a single agent for the treatment of patients with locally advanced or metastatic non-small-cell lung cancer (NSCLC) after failure of at least one prior chemotherapy regimen and in combination with gemcitabine for first line treatment of patients with locally advanced, unresectable or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects accrue to one of two phases:

  * in the Dose Escalation Phase, the subject has a histologically confirmed solid tumor that is metastatic or unresectable and is no longer responding to therapies known to prolong survival or to other standard therapies, or has disease for which no standard therapy exists or for which monotherapy with erlotinib is considered standard therapy.
  * in the Cohort Expansion Phase, the subject has advanced or metastatic NSCLC that is no longer responding to therapies known to prolong survival or to other standard therapies and which:

    1. has been previously or currently treated with erlotinib or gefitinib or
    2. with the agreement of the sponsor, has been previously or is currently treated with other EGFR/VEGFR tyrosine kinase inhibitors
* The subject has measurable or non-measurable lesions by the Response Evaluation Criteria in Solid Tumor (RECIST) criteria.
* At least 10 unstained slides of tumor tissue, archival or fresh, or paraffin block or a fresh tumor biopsy are identified and designated for central laboratory analysis.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* The subject has adequate organ and marrow function.
* The subject has a fasting plasma glucose ≤ 120 mg/dL at screening.
* The subject is ≥ 18 years old.
* The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document.
* Sexually active subjects (male and female) must use accepted methods of contraception during the course of the study and for at least 3 months after the last dose of protocol drug(s).
* Female subjects of childbearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

* The subject has previously been treated with a selective PI3K inhibitor.
* The subject has received:

  * cytotoxic chemotherapy (including investigational cytotoxic agents) or biologic agents (antibodies, immune modulators, cytokines) within 3 weeks or has received nitrosoureas or mitomycin C within 6 weeks before the scheduled first dose of XL147
  * a small-molecule kinase inhibitor (including investigational small molecule kinase inhibitors) excluding small-molecule inhibitors of EGFR or non-cytotoxic hormonal agent within 14 days of the scheduled first dose of XL147
  * other investigational therapy (ie, not specified in exclusion criterion) within 28 days of the first scheduled dose of XL147
* The subject has not recovered from toxicity due to prior therapy to baseline or Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or less (except alopecia).
* The subject has a diagnosis of uncontrolled diabetes mellitus.
* The subject is currently receiving anticoagulation with therapeutic doses of warfarin (low-dose warfarin ≤ 1mg/day, heparin, and low-molecular weight heparins are permitted).
* The subject is taking oral corticosteroids chronically.
* The subject has prothrombin time/International Normalized Ratio and/or partial thromboplastin time test results at screening that are above 1.3x the laboratory upper limit of normal.
* The subject has uncontrolled intercurrent illness including but not limited to an active infection or hypertension that would limit compliance with study requirements.
* The subject has had congestive heart failure, unstable angina, a myocardial infarction, or a stroke within 3 months of entering the study.
* The subject has a baseline corrected QT interval (QTc) ≥ 460 ms.
* The subject has psychiatric illness/social situation(s) that would limit compliance with study requirements.
* The subject is known to be positive for the human immunodeficiency virus.
* The subject has a previously identified allergy or hypersensitivity to components of the XL147 formulation.
* The subject is pregnant or breastfeeding.
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, and maximum tolerated dose of XL147 administered in combination with erlotinib | Assessed during periodic visits

SECONDARY OUTCOMES:
To evaluate plasma pharmacokinetics of XL147 and erlotinib when administered in combination | Assessed during periodic visits
To evaluate preliminary efficacy of XL147 in combination with erlotinib in adults with refractory solid tumors | Assessed during periodic visits

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 1214, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Soria JC, LoRusso P, Bahleda R, Lager J, Liu L, Jiang J, Martini JF, Mace S, Burris H. Phase I dose-escalation study of pilaralisib (SAR245408, XL147), a pan-class I PI3K inhibitor, in combination with erlotinib in patients with solid tumors. Oncologist. 2015 Mar;20(3):245-6. doi: 10.1634/theoncologist.2014-0449. Epub 2015 Feb 10. PMID 25669662